CLINICAL TRIAL: NCT06219265
Title: Neuropsychological and Electrophysiological Effects of Dance Therapy With People With Severe Mental Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asociación Canaria de Terapias Creativas (ASCATEC) (Other)
Responsible Party: Principal Investigator, Nayra Caballero Estebaranz, Director of ASCATEC and Department of Health Sciences, European University of the Canary Islands, Asociación Canaria de Terapias Creativas (ASCATEC)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TFM_01_DANZA
Record Dates: First submitted 2023-12-28; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Severe Mental Disorder
Keywords: Dance Therapy; Electroencephalography; Cognition; Severe Mental Disorder
MeSH Terms: conditions — Mental Disorders | interventions — Dance Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group 1: people with SMD receiving dance therapy (Experimental): Intervention group of people with SMD (n=26) who receive a 20-session dance therapy program for 10 weeks with 2 sessions per week in which they work for 1 hour on memory, attention and executive functions through dance and movement, ending with 10 minutes of Mindfulness.
  Interventions: Behavioral: Dance Therapy
- Control group: people with SMD who do not receive any intervention (No Intervention): This group of 21 persons with SMD will not receive any intervention.

INTERVENTIONS:
Behavioral: Dance Therapy — A single-centre prospective randomised controlled trial will be conducted with a minimum of 48 patients with severe mental disorder (SMD) who will be randomised into two groups, 1 intervention group receiving dance therapy (n=24) and 1 control group receiving no intervention or treatment (n=24).
  In addition, there will be an intervention group of healthy people who will receive dance therapy (n=20).
  All the tests, will be carried out with patients with SMD and only the EEG for healthy people, in order to determine their baseline state. The dance therapy program will last for 20 sessions over 10 weeks.
  The 44 people in the two experimental groups will participate in a 10-week intervention program with 2 sessions per week in which they will work for 1 hour on memory, attention and executive functions through dance and movement, ending with 10 minutes of Mindfulness.
  The 24 people in the control group will not receive any type of intervention.
  Arms: Experimental group 1: people with SMD receiving dance therapy

SUMMARY:
A single-centre prospective randomised controlled trial will be conducted with a minimum of 47 patients with severe mental disorder (SMD) who will be randomly assigned into two groups, 1 intervention group receiving dance therapy (n=26) and 1 control group who will not receive any intervention or added treatment apart from continuing with their usual treatment (pharmacological), but will not receive intervention with dance therapy (n=21).

In summary, the groups are:

* Experimental group (n=26): people with SMD receiving dance therapy.
* Control group (n=21): people with SMD who do not receive the dance therapy intervention but do receive their usual pharmacological treatment.

Tests will be administered before the start of the study and at the end of the study, as well as 3 months after the end of the study in order to compare the results between groups.

DETAILED DESCRIPTION:
All the tests (BASC, MoCA, PANSS and EEG) will be carried out with the 47 patients with SMD to find out their baseline status. The people with SMD will be randomly assigned to an experimental group (dance therapy program) or a control group (without intervention in dance therapy but with regular pharmacological treatment). The study will last approximately 1 year between the administration of tests, the program and the analysis of results. The dance therapy program will last 20 sessions over 10 weeks. The sessions will take place at the headquarters of the Canarian Association of Creative Therapies (ASCATEC) in the 21st century space in Santa Cruz de Tenerife.

The 26 people with SMD in the experimental group will participate in a 10-week intervention program with 2 sessions per week in which they will work for 1 hour on memory, attention and executive functions through dance and movement, ending with 10 minutes of Mindfulness.

The 21 people in the control group will not receive any type of dance therapy intervention, but will continue with their usual pharmacological treatment.

The effects will be measured after a treatment of 20 sessions (twice a week). Results will be obtained by analysing EEG parameters (EEG amplitude and frequency) and cognitive functions (BACS and MoCA). On the other hand, at the end of the 20-session programme, tests will also be administered to assess the symptomatology of the severe mental disorder suffered by the person (PANSS) to assess the effects of the program on these variables.

ELIGIBILITY:
Inclusion Criteria:

* Persons diagnosed with a serious mental disorder according to the Diagnostic and Statistical Manual of Mental Disorders -V.
* Have the capacity to decide and consent.
* Be between 18 and 75 years of age.
* No active consumption of toxic substances (except nicotine).
* Commitment to attend for the entire study period from December 2023 to December 2024.

Exclusion Criteria:

* Not having given free consent to participate in the study.
* Having a comorbid severe mental disorder, associated intellectual disability, history of severe brain damage or neurological disorder that may function as a confounding factor (Associated organic-type disorder, borderline or lower IQ)
* Active substance abuse (except nicotine)
* Having a cochlear implant, fixed hearing aids or plates in the head.
* Having suffered a concussion to the head with loss of consciousness that subsequently triggered symptoms related to the pathology.
* Having suffered from epileptic seizures.
* Not having the desire to participate in dance therapy sessions for any reason or to undergo electroencephalogram testing.
* Currently involved and participating in another cognitive rehabilitation program.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Brief Assessment of Cognition in Schizophrenia (BACS) | At baseline, up to 10 weeks of dance therapy program and 3 months after the end of the program.
  It is used to quantify cognitive impairment in schizophrenia. BACS includes assessments of verbal memory, working memory (Digit Span), motor speed (Motor Token), verbal fluency, attention and processing speed (Symbol Encoding) and executive function (Tower of London). Each item assessed has its own specific score.
  These scores are used to assess performance on each of the BACS subtests. Subsequently, a composite score is usually calculated that summarises the individual's overall cognitive performance.
Montreal Cognitive Assessment (MoCA) | At baseline, up to 10 weeks of dance therapy program and 3 months after the end of the program.
  30-question test to assess mild cognitive dysfunction by assessing executive function and visuospatial ability, identification, short-term memory, delayed recall, attention, language, abstraction, animal naming and orientation. Scores range from 0 to 30 and the cut-off point value for a normal score is >26 points. The test is administered in about 10-12 minutes.
Electroencephalogram (EEG) | At baseline, up to 10 weeks of dance therapy program and 3 months after the end of the program.
  The brain wave signals shall be recorded by a 14-channel electroencephalogram, whose electrodes (salt sensors) are arranged at positions A F 3, F7, F3, F C 5, T7, P7, O1, O2, P8, T8, F C 6, F4, F8 and A F 4, according to the international 10-20 system. The device also has 2 reference points at positions P3 and P4.

SECONDARY OUTCOMES:
Positive and Negative Symptom Scale (PANSS) | At baseline, up to 10 weeks of dance therapy program and 3 months after the end of the program.
  It monitors the progress of symptoms in severe mental disorders by means of 30 items that are grouped into three main dimensions: positive symptoms, negative symptoms and general symptoms. Each item is scored from 0 (no symptoms) to 7 (extreme severity) points.

CONTACTS AND LOCATIONS:
Overall Officials: Nayra Caballero Estebaranz, Principal Investigator — ASCATEC and European University of the Canary Islands
Locations (1):
- ASCATEC, Santa Cruz de Tenerife, Canary Islands, Spain

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT06219265/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT06219265/ICF_001.pdf